CLINICAL TRIAL: NCT02786199
Title: Histological Differentiation Grade Predicted by Ultrasound Backscatterer Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201505107RINA
Record Dates: First submitted 2016-04-05; First posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Neoplastic Disease; Pathology
Keywords: Hepatocellular Carcinoma(HCC); Ultrasound; Backscatter; Differentiation grade; Survival
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatocellular carcinoma: patients HCC who are going to receive surgical resection

SUMMARY:
Histological grade of hepatocellular carcinoma (HCC) is an important prognostic factor affecting patient survival. It has been divided into four grades from I to IV on the basis of histological differentiation. Grade I is the best differentiated consisting of small tumor cells arranged in thin trabeculae. Cells with higher grade are larger and less differentiated with hyperchromatic nuclei and loss of trabecular pattern.

Ultrasound is an imaging modality frequently used to evaluate liver tumors because of its convenience, real-time, less expensive and no radiation exposure. However, ultrasonographic evaluation by conventional B-mode image is semi quantitative and subjective. It still cannot replace liver biopsy for the evaluation of HCC.

This study is aimed to quantify the image characters of B-mode image and the scatterer properties using Nakagami distribution. Nakagami parameter is a general model to describe the distribution of scatterers. Therefore, the investigators hypothesized that Nakagami parameter may also reflect the histological changes in different grades of HCC.

In this study, the resected HCC tumor samples will be collected from the participants who are going to receive surgical resection, and the tumor US images and Nakagami values will be obtained via the single-element ultrasound system. The correlation between the ultrasound backscatter parameter and the differentiation grade will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 75
* Patients with HCC who underwent surgery
* The resected tumor was measured larger than 3 cm

Exclusion Criteria:

* Patients who have received other treatment in 6 months
* Patients who couldn't regular follow-up

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC who have received surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | within two years after surgery
  Suspected recurrences will be confirmed by CT or MRI.
Liver-related mortality | five years

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Ho, MD, Principal Investigator — Department of Surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No